CLINICAL TRIAL: NCT00001356
Title: Culture and Characteristics of Mastocytosis Mast Cells
Brief Title: Characteristics of Mast Cells in Mastocytosis
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 930136; 93-I-0136
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-05

CONDITIONS: Mastocytosis
Keywords: IL-3; Stem Cell Factor; Cytokines; Cell Differentiation; Receptors; Bone Marrow; Mastocytosis
MeSH Terms: conditions — Mastocytosis

SUMMARY:
This study will determine what growth factors are involved in promoting and inhibiting mastocytosis-an abnormal increase of mast cells in one or more organ systems. Mast cells release chemicals that can cause itching, blisters, flushing, bone pain, and abdominal pain. Little is known about the disease and there is no cure. Steroids and antihistamines can help reduce some symptoms.

Patients from birth to 80 years of age with increased mast cells in at least one organ system may be eligible for this 3-year study. Family members may also be enrolled for genetic testing.

Patients will be evaluated yearly at the NIH Clinical Center with the following tests and procedures:

* Medical history and physical examination.
* Blood samples.
* Laboratory blood tests, as medically indicated.
* Bone marrow aspiration and biopsy - For the bone marrow aspiration and biopsy, the back hipbone is punctured with a sterile needle. Five milliliters (1 teaspoon) of marrow is withdrawn through a syringe and a 1/2-inch piece of tissue is extracted with a special needle.

The blood and bone marrow samples will be used for clinical care and for research to determine if mastocytosis is due to mast cell growth factors or genetic changes.

Patients who require further evaluation and tests will have recommendations made to their primary physician. Any patient who requires immediate treatment will be admitted to the hospital. Standard medical treatment may include antihistamines for itching; steroids for severe abdominal symptoms such as cramping, diarrhea, and evidence of increased mast cells determined by an upper GI study; and adrenaline for anaphylactic shock. Patients who do not respond to conventional treatment may be offered participation in an experimental therapy study.

Participating family members will have a medical history and a blood sample drawn to look for genetic abnormalities.

DETAILED DESCRIPTION:
This protocol is designed to examine those growth potentiating and inhibiting factors which regulate mast cell number in patients with mastocytosis, and to explore the molecular basis of the disease process in hopes of improving therapy. Patients entered into the study are seen initially and may elect to be reevaluated yearly. The majority of patients to be entered into this protocol are currently followed at NIH on other protocols. Medical workup and treatment are in accordance with standard medical practice. The protocol is for 3 years, to be extended as facilities, faculty, and patients permit.

ELIGIBILITY:
Subjects include children and adults from birth to 80 years of age.

Participants must have histologic evidence of an increased mast cell number in at least one organ system.

Must be willing to be seen at the NIH according to protocol guidelines.

Routine medical care must be available through their referral physician.

Patients with mastocytosis now followed at the NIH on protocol 88-I-0190 will be continued on this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 1993-05; Study Completion 2002-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Kirshenbaum AS, Kessler SW, Goff JP, Metcalfe DD. Demonstration of the origin of human mast cells from CD34+ bone marrow progenitor cells. J Immunol. 1991 Mar 1;146(5):1410-5. PMID 1704394
- [Background] Kirshenbaum AS, Goff JP, Kessler SW, Mican JM, Zsebo KM, Metcalfe DD. Effect of IL-3 and stem cell factor on the appearance of human basophils and mast cells from CD34+ pluripotent progenitor cells. J Immunol. 1992 Feb 1;148(3):772-7. PMID 1370517
- [Background] Kettelhut BV, Metcalfe DD. Pediatric mastocytosis. J Invest Dermatol. 1991 Mar;96(3):15S-18S. PMID 1705949